CLINICAL TRIAL: NCT01890616
Title: Constipation and Gut Transit in Duchenne Muscular Dystrophy Patients
Brief Title: Constipation and Gut Transit in DMD Patients
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-1312
Record Dates: First submitted 2013-06-26; First posted 2013-07-02 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Constipation; DMD
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Motility: This arm will ingest the SmartPill.
  Interventions: Device: SmartPill ingestion

INTERVENTIONS:
Device: SmartPill ingestion — The participant would ingest the SmartPill and wear the data receiver for up to 5 days.

SUMMARY:
In this research study the investigators want to screen Duchenne Muscular Dystrophy (DMD) patients for signs and symptoms of constipation in patients over 18.

The investigators hypothesized:

* DMD patients have a high prevalence of constipation than in the general population.
* Prevalence of constipation will increase with age and with worsening functional status.

DETAILED DESCRIPTION:
The following procedures will take place during the study.

Constipation Assessment:

* The patient will be asked to complete a questionnaire about any symptoms of constipation.
* A physician from the study team will perform an abdominal physical exam
* The patient will have routine x-rays that monitor for spine compression fractures. These films will also be used to assess stool content.

Clinical Information The following information will also be collected during the clinic visit ;

* Age at diagnosis and genetic mutation
* Age at loss of ambulation if applicable
* Medications
* Functional status

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of Duchenne Muscular Dystrophy (based on clinical presentation and verified by compatible muscle biopsy or known dystrophin gene mutation).
* Age greater than or equal to 18 years old

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: DMD patients 5-18 yr of age who are seen in a large interdisciplinary DMD center.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2015-07-01 (Actual)

PRIMARY OUTCOMES:
GI transit times | up to 5 days
  Gi transit times will be computed by an investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Kaul, MD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States